CLINICAL TRIAL: NCT03726580
Title: Evaluation of Neurotoxic Effect of Sevoflurane-Based Anaesthesia Guided by Significant Short-Term Olfactory Identification Impairment in Old Age
Brief Title: Evaluation of Neurotoxic Effect of Sevoflurane-Based AnaesthesiaGuided by Short-Term Olfactory Identification
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Amer Galal Younis,MD (Unknown)
Responsible Party: Principal Investigator, Ahmed Said Elgebaly,MD, director, Tanta University
Other Study IDs: TantaF
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Neurotoxic Effect of Sevoflurane-Based Anaesthesia
Keywords: General anesthesia.; neurotoxicity,; olfaction,; olfactory identification.; sevoflurane.
MeSH Terms: conditions — Neurotoxicity Syndromes; Anosmia | interventions — Sevoflurane; Isoflurane; Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- control group: regional anesthesia
- general anesthesia(S): general anesthesia with sevoflurane
  Interventions: Drug: Sevoflurane
- general anesthesia(I): general anesthesia with isoflurane
- total intravenous anesthesia: total intravenous anesthesia with propofol.

INTERVENTIONS:
Drug: Sevoflurane — Assess the effect of isoflurane, sevoflurane, propofol and regional anesthesia on the olfactory threshold, olfactory identification and endocrine regulation of associative memory in the postoperative period in old age group.
  Other Names: Isoflurane; Propofol
  Groups: general anesthesia(S)

SUMMARY:
Nowadays there is increasing doubts about the safety of anesthesia . Anesthesiologists have to console the worried patients, who are anxious about the potential risks of anesthetic-induced brain damage, by suggesting that any detrimental effects would be "mild".Anesthetics are responsible for postoperative taste and odor defects and cognitive dysfunction.

DETAILED DESCRIPTION:
Aims: The aim of this study is to assess the effect of isoflurane, sevoflurane, propofol and regional anesthesia on the olfactory threshold, olfactory identification and endocrine regulation of associative memory in the postoperative period in old age group.

Methods: 600 patients (> 60years ) fulfilling the criteria of the American society of anesthesiologists and II status were selected for this prospective single-blinded randomized controlled study. Patients were randomized into one of four groups to receive regional anesthesia (control group), general anesthesia with sevoflurane, general anesthesia with isoflurane and total intravenous anesthesia with propofol.

Mini-Mental State Examination (MMSE), olfactory threshold, and olfactory identification were tested at 12 hours preoperatively (T0), at 3 hours postoperatively (T1) and at the time of discharge or postoperative 3 days (T2). In addition, serum melatonin levels were estimated at T0 and T1.

N-butyl alcohol was used to test the olfactory threshold and the Pocket Smell Test TM series (PSTs) was used to test olfactory identification. Data were analyzed using the one-way analysis of variance, Kruskal-Wallis or Mann-Whitney tests.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists I and II physical status
* aged from 60 to 75years
* scheduled for elective surgery with the anticipated duration of 100-120 min.
* surgical procedures included hernia repair,
* varicose vein surgery,
* incisional hernia repair,
* minor gynecological procedures,
* lower limb orthopedic procedures,
* minor urological procedures

Exclusion Criteria:

* Patients with recent airway infection,
* allergic rhinitis,
* nasal polyps,
* history of alcoholism,
* smoking,
* mental retardation,
* psychiatric illness,
* neurosurgical or oto-rhino-laryngeal surgery
* patients with a history of olfactory deficits and cognitive impairment

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Six hundred patients of both sex with inclusion following criteria: American Society of Anaesthesiologists I and II physical status aged from 60 to 75years scheduled for elective surgery with the anticipated duration of 100-120 min (surgical procedures included hernia repair, varicose vein surgery, incisional hernia repair, minor gynecological procedures, lower limb orthopedic procedures, and minor urological procedures)
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
The changes in Mini-Mental State Examination (MMSE) | basically at 12 hours preoperatively (T0), then 3 hours postoperatively (T1) and at the time of discharge or postoperative 3 days (T2)
  Cognitive function evaluated by MMSE scores. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia.
The changes in olfactory threshold | basically at 12 hours preoperatively (T0), then 3 hours postoperatively (T1) and at the time of discharge or postoperative 3 days (T2)
  Was measured using serial dilutions (10 dilutions) of 4% n-butyl alcohol in deionized water. The test consists of 10 steps. In each step, the odorant and a blank were presented to the participant. The test progressed from weaker-to-stronger concentrations of odorant. Two bottles were presented to each participant, an odorant bottle and an identical bottle filled with distilled water. The participant sniffed each one for approximately 9 s and then chose which one smelled stronger. If the participant was incorrect at one concentration, the next higher concentration was presented. When the correct choice was made, the same concentration of odorant was presented to the participant until four consecutive correct responses were given. The threshold was defined as the butyl alcohol concentration correctly chosen over water in four consecutive trials, and the corresponding number of the concentration was taken as the threshold value.
The changes in olfactory identification | basically at 12 hours preoperatively (T0), then 3 hours postoperatively (T1) and at the time of discharge or postoperative3 days (T2)
  Was assessed using the Pocket Smell TestTM series (PSTs). The test uses four booklets containing labels impregnated with odorous substances. The test is in multiple-choice format, with four written response alternatives for each odor. The odors are released when the labels are scratched. The examiner scraped each target patch and instructed participants to smell the patch and then select the name of the released odor from among four alternatives. Olfactory identification tested using the (PSTs) assessed both the recent memory and the remote memory of the patient as it contained odors which were a mixture of both the familiar and unfamiliar ones to the study population. Here, it is not utilized to identify patients with anosmia or hyposmia. Instead, the (PSTs) is used as a linear, unbiased unidimensional Rasch measure of human smell recognition abilities.

SECONDARY OUTCOMES:
The changes in olfactory melatonin levels | serum melatonin levels were estimated basically at 12 hours preoperatively (T0), then 3 hours postoperatively (T1) and at the time of discharge or postoperative3 days (T2)
  Melatonin levels were measured in plasma by the enzyme-linked immunosorbent assay (ELISA) (IBL, Hamburg, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: ahmed S Elgebaly, MD, Study Director — Tanta University
Locations (1):
- Ahmed Said Elgebaly, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Friedrich H, Caversaccio M, Landis BN. Olfactory disorders after general anesthesia. J Clin Anesth. 2013 Feb;25(1):73. doi: 10.1016/j.jclinane.2012.07.002. Epub 2012 Dec 12. No abstract available. PMID 23246491
- [Result] Shen X, Liu Y, Xu S, Zhao Q, Guo X, Shen R, Wang F. Early life exposure to sevoflurane impairs adulthood spatial memory in the rat. Neurotoxicology. 2013 Dec;39:45-56. doi: 10.1016/j.neuro.2013.08.007. Epub 2013 Aug 27. PMID 23994303
- [Result] Saravanan B, Kundra P, Mishra SK, Surianarayanan G, Parida PK. Effect of anaesthetic agents on olfactory threshold and identification - A single blinded randomised controlled study. Indian J Anaesth. 2018 Aug;62(8):592-598. doi: 10.4103/ija.IJA_245_18. PMID 30166653
- [Result] Obayashi K, Saeki K, Iwamoto J, Tone N, Tanaka K, Kataoka H, Morikawa M, Kurumatani N. Physiological Levels of Melatonin Relate to Cognitive Function and Depressive Symptoms: The HEIJO-KYO Cohort. J Clin Endocrinol Metab. 2015 Aug;100(8):3090-6. doi: 10.1210/jc.2015-1859. Epub 2015 Jun 8. PMID 26052727
- [Result] Kalsbeek A, Cutrera RA, Van Heerikhuize JJ, Van Der Vliet J, Buijs RM. GABA release from suprachiasmatic nucleus terminals is necessary for the light-induced inhibition of nocturnal melatonin release in the rat. Neuroscience. 1999;91(2):453-61. doi: 10.1016/s0306-4522(98)00635-6. PMID 10366002
- [Result] Lehrner JP, Gluck J, Laska M. Odor identification, consistency of label use, olfactory threshold and their relationships to odor memory over the human lifespan. Chem Senses. 1999 Jun;24(3):337-46. doi: 10.1093/chemse/24.3.337. PMID 10400452
- [Result] Rawal S, Hoffman HJ, Honda M, Huedo-Medin TB, Duffy VB. The Taste and Smell Protocol in the 2011-2014 US National Health and Nutrition Examination Survey (NHANES): Test-Retest Reliability and Validity Testing. Chemosens Percept. 2015 Sep;8(3):138-148. doi: 10.1007/s12078-015-9194-7. Epub 2015 Aug 7. PMID 27833669
- [Result] Jackman AH, Doty RL. Utility of a three-item smell identification test in detecting olfactory dysfunction. Laryngoscope. 2005 Dec;115(12):2209-12. doi: 10.1097/01.mlg.0000183194.17484.bb. PMID 16369168
- [Result] Kostopanagiotou G, Kalimeris K, Kesidis K, Matsota P, Dima C, Economou M, Papageorgiou C. Sevoflurane impairs post-operative olfactory memory but preserves olfactory function. Eur J Anaesthesiol. 2011 Jan;28(1):63-8. doi: 10.1097/EJA.0b013e328340702b. PMID 20962652
- [Result] Lotsch J, Reichmann H, Hummel T. Different odor tests contribute differently to the evaluation of olfactory loss. Chem Senses. 2008 Jan;33(1):17-21. doi: 10.1093/chemse/bjm058. Epub 2007 Aug 30. PMID 17761724
- [Result] Lecker I, Yin Y, Wang DS, Orser BA. Potentiation of GABAA receptor activity by volatile anaesthetics is reduced by alpha5GABAA receptor-preferring inverse agonists. Br J Anaesth. 2013 Jun;110 Suppl 1(Suppl 1):i73-81. doi: 10.1093/bja/aet038. Epub 2013 Mar 27. PMID 23535829
- [Result] Ren Y, Zhang FJ, Xue QS, Zhao X, Yu BW. Bilateral inhibition of gamma-aminobutyric acid type A receptor function within the basolateral amygdala blocked propofol-induced amnesia and activity-regulated cytoskeletal protein expression inhibition in the hippocampus. Anesthesiology. 2008 Nov;109(5):775-81. doi: 10.1097/ALN.0b013e31818a37c4. PMID 18946287
- [Result] Salmi E, Kaisti KK, Metsahonkala L, Oikonen V, Aalto S, Nagren K, Hinkka S, Hietala J, Korpi ER, Scheinin H. Sevoflurane and propofol increase 11C-flumazenil binding to gamma-aminobutyric acidA receptors in humans. Anesth Analg. 2004 Nov;99(5):1420-1426. doi: 10.1213/01.ANE.0000135409.81842.31. PMID 15502041
- [Result] Alkire MT, Gorski LA. Relative amnesic potency of five inhalational anesthetics follows the Meyer-Overton rule. Anesthesiology. 2004 Aug;101(2):417-29. doi: 10.1097/00000542-200408000-00023. PMID 15277925
- [Result] Shen FY, Song YC, Guo F, Xu ZD, Li Q, Zhang B, Ma YQ, Zhang YQ, Lin R, Li Y, Liu ZQ. Cognitive Impairment and Endoplasmic Reticulum Stress Induced by Repeated Short-Term Sevoflurane Exposure in Early Life of Rats. Front Psychiatry. 2018 Aug 2;9:332. doi: 10.3389/fpsyt.2018.00332. eCollection 2018. PMID 30116207